CLINICAL TRIAL: NCT03449069
Title: A Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Fistulizing Crohn's Disease: Pediatric Sub-study
Brief Title: Pediatric MSC-AFP Sub-study for Crohn's Fistula
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael C. Stephens, Sponsor-Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-010539
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fistula in Ano; Crohn Disease
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSC-AFP (Experimental): This is a single treatment group study. All patients will receive treatment of a stem cell coated fistula plug.
  Interventions: Drug: MSC-AFP

INTERVENTIONS:
Drug: MSC-AFP — Patients will have a mesenchymal stromal cell coated anal fistula plug placed in their Crohn's perianal fistula tract.
  Other Names: mesenchymal stromal cell coated anal fistula plug

SUMMARY:
The purpose of this study is to determine the safety of using an autologous mesenchymal stromal cell (MSC) coated fistula plug in people with fistulizing Crohn's disease. Autologous means these cells to coat the plug come from the patient.

DETAILED DESCRIPTION:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore Bio-A Fistula Plug) in a Phase I study using a single dose of 20 million cells. 5 patients (age 12 to 17 years) with Crohn's perianal fistulas will be enrolled.

Subjects will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore fistula plug as per current clinical practice. The subjects will be subsequently followed for fistula response and closure for 24 months. This is an autologous product derived from the patient and used only for the same patient.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 12-17 years of age.
2. Residents of the United States.
3. Crohn's disease with single or multiple draining complex perianal fistulae (definition as below) for at least three months despite standard therapy (definition below).
4. Concurrent therapies with corticosteroids, 5-aminosalicylate (5-ASA) drugs, thiopurines, methotrexate (MTX), antibiotics, and anti-tumor necrosis factor (TNF) therapy are permitted.
5. All patients should have undergone a colonoscopy in last 12 months to rule out malignant or premalignant condition
6. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
7. Ability to comply with protocol
8. Competent and able to provide written informed consent (and assent where appropriate).
9. Must have failed standard medical therapy including anti-TNF agents

Exclusion Criteria

1. Inability to obtain informed consent (and assent where appropriate).
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. sepsis, pneumonia active serious infection or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions;

   a. Evidence of hepatitis B, C, or HIV
4. History of cancer including melanoma (with the exception of localized skin cancers)
5. Investigational drug within thirty (30) days of baseline
6. A resident outside the United States
7. Pregnant or trying to become pregnant, or breast feeding.
8. History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
9. Previous allergic reaction to a perianal fistula plug.
10. If adipose tissue is not technically feasible
11. Weight less than 35 kg
12. Allergic to local anesthetics
13. Non-enterocutaneous tracts (i.e. recto-vaginal, entero-vesicular)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (safety and toxicity) | 2 months to approximately at 24 months
  Participants will have a health assessment and blood work done at each study visit to monitor for adverse events.

SECONDARY OUTCOMES:
Number of participants with response to the treatment regarding cessation of drainage from the treated fistula. | 2 months to approximately at 24 months
  Participants will have a clinical assessment of fistula drainage at each study visit.
Number of participants with radiographic response to the treatment regarding the treated fistula. | Week 2, Week 8, and Week 24
  Participants will have an assessment of healing radiographically by magnetic resonance imaging (MRI) at Week 2 visit, Week 8, and Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stephens, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials